CLINICAL TRIAL: NCT06503796
Title: Antiviral Therapy in Infants With HBV Infection
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2023-12-85-1
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: HBV
MeSH Terms: interventions — Lamivudine; Interferons

STUDY DESIGN:
Intervention Model Description: the antiviral group and the control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the antiviral group (Experimental): HBV-infected infants in the treatment group were treated with LAM (4 mg/kg/d) before 1 year of age, and then combined with regular interferon (intramuscular or subcutaneous injection, 3-6 million U/m2 body surface area, every other day, with a starting dose of 3 million U/m2 body surface area, which was adjusted according to the specific tolerances of the children during the course of the treatment) if they were still HBV DNA and/or HBsAg-positive at the end of the 1st year of age. The course of interferon treatment is 52 weeks.
  Interventions: Drug: Lamivudine; Drug: Interferon
- the control group (No Intervention): synchronized follow-up visits without intervention

INTERVENTIONS:
Drug: Lamivudine — 4mg/kg/d, oral
  Arms: the antiviral group
Drug: Interferon — Use only in children who remain positive for HBV-DNA and/or HBsAg after 1 year of age. Regular interferon (3 million U/m2 body surface area, intramuscular or subcutaneous, every other day, adjusted during treatment according to the child's specific tolerance) for 52 weeks.
  Arms: the antiviral group

SUMMARY:
This study was a multicenter, prospective randomized controlled clinical study. A total of 60 HBV-infected infants with ALT ≤5 times the upper limit of normal (ULN) and without pathological jaundice were enrolled and randomized 1:1 into two groups: the control group and the antiviral treatment group. HBV-infected infants in the treatment group were treated with LAM before the age of 1 year and then combined with regular interferon for 52 weeks if they were still positive for HBV DNA and/or HBsAg after reaching the age of 1 year. The control group was followed up synchronously. Follow-up was conducted every 3 months during the study period. The main efficacy evaluation indexes: HBsAg conversion (functional cure) rate, HBeAg conversion rate, HBeAg seroconversion rate, HBV DNA conversion rate, HBsAg seroconversion rate, and ALT reversion rate at the end of 12 months of treatment and at 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* a. Age ≤ 1 year;
* b. HBsAg and HBV DNA positive;
* c. ALT ≤ 5 times the upper limit of normal (ULN) and no pathologic jaundice (two consecutive tests with an interval of 2 weeks - 3 months).
* d. Parents are willing to participate in the study and sign an informed consent form, for children without parents, all legal guardians of need to give informed consent.

Exclusion Criteria:

* a. Combined viral infections such as HAV, HCV, HDV, HEV, HIV, EBV, CMV, etc;
* b. Combination of other liver diseases, such as autoimmune hepatitis, drug-induced liver injury, Wilson's disease;
* c. WBC <9 × 10^9/L, or PLT <90 × 10^9/L;
* d. Combination of other systemic serious diseases or hereditary diseases, etc;
* e. Other conditions deemed by the investigator to be unsuitable for participation in this study.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The rate of HBsAg loss | 12months after intervention, 2 years old
  The rate of HBsAg loss in 12months after intervention, 2 years old

SECONDARY OUTCOMES:
The rate of HBsAg seroconversion | 12months after intervention, 2 years old
  The rate of HBsAg seroconversion in 12months after intervention, 2 years old
The rate of HBV DNA loss | 12months after intervention, 2 years old
  The rate of HBV DNA loss in 12months after intervention, 2 years old
The rate of HBeAg loss | 12months after intervention, 2 years old
  The rate of HBeAg loss in 12months after intervention, 2 years old
The rate of HBeAg seroconversion | 12months after intervention, 2 years old
  The rate of HBeAg seroconversion in 12months after intervention, 2 years old
ALT reversion rate | 12months after intervention, 2 years old
  ALT reversion rate in 12months after intervention, 2 years old
Incidence of Treatment-Emergent Adverse Events | 12months after intervention, 2 years old
  Safety and Tolerability of Antiviral Therapy in infants

CONTACTS AND LOCATIONS:
Overall Officials: Junliang Fu, Principal Investigator — The fifth medical center of PLA
Locations (1):
- the Fifth Medical Center of PLA, Beijing, China

IPD SHARING:
Plan to Share IPD: No